CLINICAL TRIAL: NCT03237000
Title: Effect of Administering Intravenous Magnesium Sulfate Heptahydrate (MgSO4•7H2O) on Fetal Cardiotocography and Neonatal Outcome in Preeclamptic Patients in 3rd Trimester of Pregnancy
Brief Title: Effect of Administering Intravenous Magnesium Sulfate on Fetal Cardiotocography and Neonatal Outcome in Preeclamptic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 7
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; MgSO4
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: Magnesium sulphate was administered by continuous intravenous infusion according to our hospital protocol as follows:
  * Loading dose: 4-6 gm of magnesium sulphate diluted in 100 mL of IV fluid administered over 15-20 min.
  * Maintenance dose: 2 gm/hr in 100 mL of IV infusion to be continued for 24 hours after delivery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MgSO4 (Experimental): Magnesium sulphate was administered by continuous intravenous infusion according to our hospital protocol as follows:
  * Loading dose: 4-6 gm of magnesium sulphate diluted in 100 mL of IV fluid administered over 15-20 min.
  * Maintenance dose: 2 gm/hr in 100 mL of IV infusion to be continued for 24 hours after delivery.
  Interventions: Drug: MgSO4

INTERVENTIONS:
Drug: MgSO4 — Magnesium sulphate was administered by continuous intravenous infusion according to our hospital protocol as follows:
  * Loading dose: 4-6 gm of magnesium sulphate diluted in 100 mL of IV fluid administered over 15-20 min.
  * Maintenance dose: 2 gm/hr in 100 mL of IV infusion to be continued for 24 hours after delivery.
  Other Names: Magnisium sulfate

SUMMARY:
Admission CTG for 20 minutes Settings on a CTG machine was standardised to enable a consistent approach of interpretation of traces. Paper speed of 3cm per minute will be adopted. Maternal heart rate was recorded and noted on CTG. Following birth date, time and mode of delivery will be labelled on CTG.

Magnesium sulphate was administered by continuous intravenous infusion according to our hospital protocol as follows:

* Loading dose: 4-6 gm of magnesium sulphate diluted in 100 mL of IV fluid administered over 15-20 min.
* Maintenance dose: 2 gm/hr in 100 mL of IV infusion to be continued for 24 hours after delivery.

Another 20 minutes CTG strip will be performed 20 minutes after administration of IV loading MgSO4, 7H2O and thus ensuring that MgSO4 has reached peak serum levels

DETAILED DESCRIPTION:
Admission CTG:

Admission CTG will be performed for 20 minutes

I-Settings:

1. Settings on a CTG machine will be standardised to enable a consistent approach of interpretation of traces.
2. Paper speed of 3cm per minute will be adopted.
3. CTGs will be labelled with mother's name, hospital number.
4. Date and time settings on machines will be labelled at commencement of tracing.
5. Maternal heart rate will be recorded and noted on CTG.
6. Following birth date, time and mode of delivery will be labelled on CTG.

Magnesium Sulphate hepatahydrate administration:

Magnesium sulphate will be administered by continuous intravenous infusion according to our hospital protocol as follows:

* Loading dose: 4-6 gm of magnesium sulphate diluted in 100 mL of IV fluid administered over 15-20 min.
* Maintenance dose: 2 gm/hr in 100 mL of IV infusion to be continued for 24 hours after delivery.
* Magnesium toxicity was monitored by hourly assessment of:

  1. Patellar reflexes should be present.
  2. Respiratory rate not < 16/min.
  3. Urine output not < 100ml / hr. Another 20 minutes CTG strip will be performed 20 minutes after administration of IV loading MgSO4, 7H2O and thus ensuring that MgSO4 has reached peak serum levels

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant Women in the third trimester.
2. Severely preeclamptic patients.
3. Singleton Pregnancy.
4. Patients with normal admission CTG

Exclusion Criteria:

1. Evidence of fetal anomalies on scan.
2. Concomitant maternal morbidities as diabetes, cardiac disease.
3. Patients contraindicated to take MgSo4 e.g.: advanced renal disease.
4. Abnormal admission CTG.
5. Morbid obesity.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Fetal heart rate tracing | 20 minutes after MgSO4 administration
  Settings on a CTG machine is standardised to enable a consistent approach of interpretation of traces. Paper speed of 3cm per minute is adopted

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt